CLINICAL TRIAL: NCT00006381
Title: Phase II Study of Celecoxib in HER-2/Neu Overexpressing Metastatic Breast Cancer Patients Who Have Failed Recombinant Humanized Anti-p 185HER Monoclonal Antibody Trastuzumab (HERCEPTIN)
Brief Title: Celecoxib and Trastuzumab in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068255; MSKCC-00078; NCI-G00-1869
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2003-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Celecoxib

INTERVENTIONS:
Biological: trastuzumab
Drug: celecoxib

SUMMARY:
RATIONALE: Celecoxib may be effective in preventing the further development of cancer. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining trastuzumab with celecoxib may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining celecoxib and trastuzumab in treating women who have metastatic breast cancer that has not responded to previous trastuzumab.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of celecoxib and trastuzumab (Herceptin) in women with HER2/neu-overexpressing metastatic breast cancer that is refractory to prior trastuzumab.
* Determine the safety of celecoxib in these patients.

OUTLINE: At least 3 weeks after the last dose of prior chemotherapy, patients receive oral celecoxib twice daily. Patients continue or restart trastuzumab (Herceptin) IV over 30-90 minutes weekly or every 3 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within approximately 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic breast cancer

  * HER2/neu-positive (overexpressing) tumor tissue
* Failed prior trastuzumab (Herceptin) therapy with or without chemotherapy
* Resected stage IV disease allowed if evidence of disease
* Bidimensionally measurable or evaluable disease

  * No lesions in previously irradiated field except nonbone lesions progressive after radiotherapy
  * No pleural effusions
  * No blastic or mixed bony metastases
  * No palpable abdominal masses
* No leptomeningeal disease
* Brain metastases allowed if:

  * No concurrent use of steroids
  * At least 3 months since prior brain irradiation
  * No evidence of progression of metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Hemoglobin at least 8.0 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* AST/ALT no greater than 2 times upper limit of normal (ULN)
* Bilirubin no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* LVEF at least 50%

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No other prior malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No other serious medical illness
* No severe infection
* No severe malnutrition
* No prior allergic reactions to sulfonamides or celecoxib

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* Prior trastuzumab (Herceptin) for breast cancer allowed, either as adjuvant/neoadjuvant or for metastatic disease

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior cytotoxic therapy for breast cancer allowed, either as adjuvant/neoadjuvant or for metastatic disease

Endocrine therapy:

* See Disease Characteristics
* At least 3 weeks since prior hormonal therapy
* Prior exogenous hormonal therapy for stage IV disease and/or as adjuvant therapy allowed

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* Prior localized radiotherapy allowed if no influence on the signal measurable lesion
* Concurrent localized radiotherapy allowed if no influence on the signal measurable lesion

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior major surgery and recovered
* At least 2 weeks since prior minor surgery and recovered

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chau T. Dang, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States